CLINICAL TRIAL: NCT07087145
Title: Persistent Oral HPV Among Diverse PLWH: A Pilot Study to Evaluate the Feasibility and Acceptability of Testing for Oral HPV DNA Infection With Mail-delivered Sample Collection Kits
Brief Title: Feasibility of HPV Testing With Mail-delivered Sample Collection Kits
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 240514; R03DE033930 (NIH)
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: HPV Infection; HIV Infections; HPV-Related Malignancy
Keywords: HPV Testing
MeSH Terms: conditions — Papillomavirus Infections; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Three saliva samples will be collected for analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Samples from Persons Living With HIV (PLWH): Participants will complete an online survey and receive a sample collection kit in the United States (US) mail. Two saliva samples will be obtained at home (one sample collected with two foam swabs and applied to a single FTA indicating card) and one oral rinse and gargle sample. Participants will complete a follow-up survey, and 7-10 days after the date of home sample collection, participants will visit the UCSF Anal Neoplasia Clinic, Research and Education (ANCRE) Clinic at Mt. Zion for a 15-minute clinic visit. During this clinic visit, participants will additionally complete one oral rinse and gargle sample.
  Interventions: Diagnostic Test: Mail-based Saliva Sample Kit; Other: Study-related Surveys

INTERVENTIONS:
Diagnostic Test: Mail-based Saliva Sample Kit — Sent via United States Postal Service and returned via FedEx
  Other Names: Mail-based Specimen Sample Kit
Other: Study-related Surveys — Online surveys will be administered
  Other Names: Web-based Surveys

SUMMARY:
People living with human immunodeficiency virus (PLWH) have an estimated 1.6-6.0 times increased risk of developing oropharyngeal cancer (OPC) compared with individuals in the general population. 70% of OPCs are caused by human papillomavirus (HPV), and PLWH also have an increased prevalence of oral HPV infection. Disparities by race/ethnicity also include a later stage of diagnosis and less frequent cancer-directed treatment for members of ethnic minority groups. There is little known regarding the racial/ethnic differences in oral HPV infection, persistence of oral HPV infection, or progression of oral HPV infection to OPC among PLWH. This is an observational, prospective cohort study to investigate the feasibility of alternative sample collection methods for HPV testing among PLWH.

DETAILED DESCRIPTION:
STUDY AIMS:

1. To determine if oral HPV deoxyribonucleic acid (HPV DNA) results obtained from self-collected oral rinse and gargle samples (ORG) sent by mail agree with results obtained from ORG samples collected in a clinic setting, among race/ethnically diverse sexual minority men (SMM) living with HIV (LWH).
2. To determine if oral HPV DNA results obtained from self-collected saliva samples applied to a Flinders Technology Associates (FTA) card sent by mail agree with results obtained from (1) ORG samples collected in a clinic setting, and (2) Home ORG, among race/ethnically diverse SMM-LWH.
3. To determine the feasibility, acceptability, and comfort of receiving HPV DNA sample collection kits by mail, self-collecting samples, and returning samples by FedEx, among racially/ethnically diverse SMM-LWH.

OUTLINE:

Participants will provide two saliva samples (at the same time), complete surveys, and complete a single clinic visit. Follow-up will be between 7 and 10 days post initial sample collection.

ELIGIBILITY:
Inclusion Criteria:

1. Over 35 years of age
2. Member of a sexual or gender group considered sexual minority men (men who have sex with men, trans-women)
3. Person living with HIV
4. Willing and able to receive a package through United States (US) postal service
5. Willing and able to return a package through FedEx
6. Able to attend a clinic visit at University of California, San Francisco (UCSF) Mt. Zion campus

Exclusion Criteria:

* Does not meet the above criteria

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults living with HIV (PLWH)
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2024-11-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with positive oral human papillomavirus infection | Up to 10 days
  The prevalence of oral high-risk human papillomavirus (hrHPV) infection will be determined by the percentage of participants with a positive result for human papillomavirus deoxyribonucleic acid (HPV DNA) after testing
Agreement in the detection of oral HPV DNA between the oral rinse and gargle (ORG) and the clinic sample | Up to 10 days
  The agreement in the detection of oral HPV DNA between the oral rinse and gargle (ORG) sample collected at home and the sample collected at the clinic will be measured using kappa. The Kappa Coefficient, often denoted as κ (kappa), is a statistical measure used to assess the level of agreement between two events providing a way to quantify the extent to which the observed agreement exceeds what would be expected by chance alone. The Kappa Coefficient ranges from -1 to 1, where 1 indicates perfect agreement, 0 indicates no agreement beyond chance, and negative values suggest less agreement than would be expected by random chance. Substantial agreement is considered kappa (κ) at least ≥0.61
Agreement in the detection of oral HPV DNA between Flinders Technology Associates (FTA) sample collection card and both the ORG samples (Home and Clinic). | Up to 10 days
  The agreement in the detection of oral HPV DNA between the sample collected and applied to an FTA sample collection card (FTA) and both the ORG samples (Home and Clinic). will be measured using kappa. The Kappa Coefficient, often denoted as κ (kappa), is a statistical measure used to assess the level of agreement between two events providing a way to quantify the extent to which the observed agreement exceeds what would be expected by chance alone. The Kappa Coefficient ranges from -1 to 1, where 1 indicates perfect agreement, 0 indicates no agreement beyond chance, and negative values suggest less agreement than would be expected by random chance. Substantial agreement is considered kappa (κ) at least ≥0.61

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Hernandez Levenston, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No